CLINICAL TRIAL: NCT01144221
Title: Protocol on an Evaluative Study on Bone Marrow Derived Mononuclear Cells for Optimization of Biventricular Pacing in Patients With Chronic Ischemic Left Ventricular Dysfunction
Brief Title: Bone Marrow Derived Mononuclear Cells for Ischemic Cardiomyopathy
Acronym: Alster-Star
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: funding issues
Sponsor: Kai Jaquet, PhD, DSc (Industry)
Responsible Party: Sponsor-Investigator, Kai Jaquet, PhD, DSc, Head of Stem Cell Lab, Asklepios proresearch
Organization: Asklepios proresearch (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1764; 2008-008368-28 (EudraCT Number)
Record Dates: First submitted 2010-06-14; First posted 2010-06-15 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2012-08

CONDITIONS: Heart Disease
Keywords: Chronic Ischemic Heart Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stem cell treatment (Experimental): Patients treated via stem cell injection
  Interventions: Procedure: Intramyocardial Cell therapy

INTERVENTIONS:
Procedure: Intramyocardial Cell therapy — Intramyocardial Cell therapy in patients with chronic ischemic heart disease after ICD CRT Implantation

SUMMARY:
This is an evaluative, monocentric study in patients with chronic ischemic heart disease and left bundle branch block who received an ICD-CRT. It is an early investigation on the safety and effects of a single administration of bone marrow derived mononuclear cells after implantation of an ICD-CRT device as an adjunct to CRT and usual drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* chronic left ventricular dysfunction (ejection fraction <35 %) in chronic ischemic heart disease and asynchronic contraction with indication for a biventricular stimulation (CRT, chronic resynchronization therapy), who do not have an improvement of >15% of LVEF 3 months after CRT-device implantation
* wall motion dysfunction of any territory
* left bundle branch block
* Patients were on individual optimal treatment for chronic ischemic heart disease with one or a combination of the following drug types: diuretics, ß-blockers, ACE-inhibitors, AT1 blockers and/or lipid lowering agents for at least 30 days before CRT Implantation

Exclusion Criteria:

* patients with left ventricular dysfunction due to other reasons than ischemic cardiomyopathy, e.g. hypertension, dilatative cardiomyopathy
* with relevant valvular disease;
* Aneurysma of the anterior myocardial wall or myocardial wall thickness of < 5 mm,
* with overt heart failure, other than ischemic cardiomyopathy,
* with history of stroke and/or transient ischemic attack (TIA),
* with history of thromboembolic event (e.g. phlebothrombosis, pulmonary embolism), bleeding disorders and known disease of the coagulation system;
* with extensive deviations of baseline laboratory values and significant findings at physical examination which in the opinion of the investigator may worsen under treatment;
* with severe systemic disease - (e.g. known or suspected anaphylaxia, intolerance against X-ray or contrast agent and, pre-malignant and malignant disease)
* atrial fibrillation with average heart rate >70 bpm
* pregnant women and women of childbearing potential who have not had a negative pregnancy test within 48 hours before treatment;
* with any disease or condition that seriously compromises the function of other body systems than the heart and/or might interfere with conduct of the study and interpretation of the results;
* patients with a chronic or acute HIV-, HBV-, HCV-infection;
* improvement of more than 15% of LVEF 3 months after CRT-device implantation
* patients who have a ICD Implantation for secondary prophylactic indication. These patients show a history of resuscitation, VT or syncope.
* patients who are currently participating in another investigational drug or device study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
LVEF Value | 12 months
  LVEF values will be compared after ICD CRT-Implantation and after Bone Marrow Derived Mononuclear Cells Injection

CONTACTS AND LOCATIONS:
Overall Officials: Korff Krause, Dr. med., Principal Investigator — Asklepios proresearch
Locations (1):
- Asklepios Clinic St. Georg, Hamburg, Germany